CLINICAL TRIAL: NCT01567124
Title: A Randomised Trial Examining the Effectiveness of Sympathetic Nervous Inhibition in Alleviating the Metabolic Side Effects of Antipsychotic Medications in Patients With Schizophrenia
Brief Title: Alleviating the Metabolic Side Effects of Antipsychotic Medications
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Collaborators: The Alfred (Other); Monash Medical Centre (Other); Ballarat Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 108/12; 1022794 (Other Grant/Funding Number: NHMRC)
Record Dates: First submitted 2012-03-25; First posted 2012-03-30 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Moxonidine; Sympathetic nervous system activation; Cardiometabolic side effects of antipsychotics
MeSH Terms: conditions — Schizophrenia | interventions — moxonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olanzapine (Other): Participants taking olanzapine at the time of recruitment will continue to take this medication as part of standard care for schizophrenia.
  Interventions: Drug: Moxonidine; Drug: Placebo
- Clozapine (Other): Participants taking clozapine at the time of recruitment will continue to take this medication as part of standard care for schizophrenia.
  Interventions: Drug: Moxonidine; Drug: Placebo

INTERVENTIONS:
Drug: Moxonidine — Participants who are randomly assigned to the moxonidine/experimental group will be treated with moxonidine oral tablets for twelve weeks. Participants will begin their moxonidine treatment at 0.2mg dosage, which will be increased to 0.4mg over the first two weeks.
  At the end of the twelve weeks of treatment, participants will be withdrawn from moxonidine over a period of two weeks.
  Other Names: Physiotens
  Arms: Olanzapine
Drug: Placebo — To examine the effects of moxonidine treatment, a placebo oral tablet will be used for comparison purposes.
  The duration and number of placebo tablets participants will be required to take will be the same as the amount required in the moxonidine group.
  Arms: Olanzapine
Drug: Moxonidine — Participants who are randomly assigned to the moxonidine/experimental group will be treated with moxonidine oral tablets for twelve weeks. Participants will begin their moxonidine treatment at 0.2mg dosage, which will be increased to 0.4mg over the first two weeks.
  At the end of the twelve weeks of treatment, participants will be withdrawn from moxonidine over a period of two weeks.
  Other Names: Physiotens
  Arms: Clozapine
Drug: Placebo — To examine the effects of moxonidine treatment, a placebo oral tablet will be used for comparison purposes.
  The duration and number of placebo tablets participants will be required to take will be the same as the amount required in the moxonidine group.
  Arms: Clozapine

SUMMARY:
The use of antipsychotic medications has increased over the past decade. While more recently developed medications are improved with regards to extrapyramidal side effects, the use of atypical antipsychotics has been associated with substantial weight gain and a worsening of metabolic profile. The time course and extent of weight gain differs among antipsychotics, with olanzapine and clozapine being associated with greatest weight gain.

Mechanisms underlying a worsening metabolic profile, obesity and obesity-related illnesses are complex, extending beyond sedentary lifestyle, poor diet and genetic predisposition. There is also a growing body of evidence that the sympathetic nervous system (SNS) has a role in the generation of both obesity and obesity-related illness. While the role of the SNS in blood pressure control is readily acknowledged it is less well appreciated that activation of the SNS exerts profound metabolic effects.

Although the fact of a causal relation linking antipsychotic drugs and obesity is unequivocally established, the biological mechanisms operating are unclear, and strategies for preventive therapy remain largely unformulated.

This study aims to investigate the role of the SNS and its association with the metabolic abnormalities that are frequently observed in patients with schizophrenia following treatment with antipsychotic medications.

Additionally, the study will investigate whether treatment with the centrally acting sympatholytic agent moxonidine will modify SNS activity and, hence, favourably influence the downstream metabolic abnormalities seen in antipsychotic treated patients with schizophrenia.

Hypothesis 1: Elevated sympathetic nervous system activity underlies the metabolic disturbances observed in patients following antipsychotic therapy.

Aim 1: To investigate the role of the sympathetic nervous system and its association with the metabolic abnormalities that are frequently observed in patients with schizophrenia following treatment with antipsychotic medications

Hypothesis 2: Central sympathoinhibition with moxonidine will blunt the elevated sympathetic nervous activity and downstream metabolic abnormalities observed in antipsychotic treated patients with schizophrenia.

Aim 2: Determine whether treatment with the centrally acting sympatholytic agent moxonidine will modify sympathetic nervous system activity and, hence, favourably influence the downstream metabolic abnormalities seen in antipsychotic treated patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years.
* Capable of understanding and willing to provide signed and dated written, voluntary informed consent in advance of any protocol-specific procedures.
* Psychiatrist confirmed diagnosis of schizophrenia.
* Stabilised on clozapine or olanzapine for at least 6 weeks.
* 5% increase in body weight since commencement of clozapine or olanzapine.

Exclusion Criteria:

* Aged < 18 or > 65 years.
* On a Community Treatment Order (CTO).
* Comorbid mental health conditions including schizoaffective disorder, personality disorders, eating disorders, mental retardation, pervasive developmental disorder, delirium, dementia (ie, Mini Mental State Examination [MMSE] < 23), and amnesia.
* Concurrent treatment with two or more antipsychotics (including clozapine or olanzapine) at screening.
* Concomitant treatment with sedatives, tricyclic antidepressants, metformin, insulin or beta adrenergic blocking agents.
* Known or suspected hypersensitivity to moxonidine.
* Previous history of clozapine induced myocarditis.
* Pre-existing and/or current diagnosed heart disease.
* Comorbid medical conditions including medicated hypertension, bradycardia (heart rate < 50 beats/min), type 1 diabetes, epilepsy, bleeding disorders, alcohol/drug dependence, infectious blood diseases, and moderate-severe renal impairment.
* Clinically significant abnormalities on examination or laboratory testing, and clinically significant medical conditions not listed above that are serious and/or unstable.
* Pregnant or breastfeeding women.
* Women of childbearing potential (WOCP) who are not using medically accepted contraception (ie, intrauterine devices [IUDs], hormonal contraceptives [oral, depot, patch or injectable], and double barrier methods such as condoms or diaphragms with spermicidal gel or foam. Women who are postmenopausal (ie, amenorrhea for at least 12 consecutive months) or surgically sterile are not considered to be WOCP.
* Sexually active men with WOCP partners who are not using medically accepted contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05

PRIMARY OUTCOMES:
To determine the association between sympathetic nervous system and metabolic abnormalities (eg, weight gain) observed with antipsychotic treatment. | Baseline and following 12 weeks of moxonidine/placebo treatment.
  To investigate the role of the sympathetic nervous system and it's association with the metabolic abnormalities that are frequently observed in patients with schizophrenia who are treated with antipsychotic medications; namely clozapine and olanzapine.

SECONDARY OUTCOMES:
Change from baseline in sympathetic nervous system activity. | Baseline and following 12 weeks of moxonidine/placebo treatment.
  We will explore whether treatment with the centrally acting sympatholytic agent, moxonidine, modifies sympathetic nervous system activity and hence, has a favourable influence on the downstream metabolic abnormalities seen in schizophrenic patients treated with antipsychotics.

CONTACTS AND LOCATIONS:
Overall Officials: Gavin Lambert, Study Director — Baker IDI Heart & Diabetes Institute; David Barton, Principal Investigator — Monash Medical Centre; Abdul Khalid, Principal Investigator — Ballarat Health Services
Locations (4):
- Australia (4):
  - Ballarat Health Service Psychiatric Services, Ballarat, Victoria
  - Monash Medical Centre - Monash Health, Clayton, Victoria
  - Alfred and Baker Medical Unit - Alfred Hospital, Melbourne, Victoria
  - Baker IDI Heart & Diabetes Institute, Melbourne, Victoria